CLINICAL TRIAL: NCT07105657
Title: The Outcome of Three Weeks Rehabilitation in Patients With a Total Hip or Knee Replacement Experiencing Persistent Physical Impairments
Acronym: Rehab-hip-knee
Status: Recruiting | Type: Observational
Sponsor: Horsens Hospital (Other)
Collaborators: VIA University College (Other)
Responsible Party: Principal Investigator, Jeppe Lange, Ass. prof., Horsens Hospital
Other Study IDs: 1-16-02-329-25
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Hip Osteoarthritis; Knee Osteoarthristis
Keywords: total hip replacement; rehabilitation; hip osteoartritis; knee osteoarthritis; total knee replacement
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention group hip: Patients with a total hip replacement undergoing rehabilitation
  Interventions: Other: Rehabilitation
- Intervention group knee: Patients with a total hip replacement undergoing rehabilitation
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — Three weeks intensive rehabilitation where patients undergo group-based and individualised rehabilitation focusing at improving pain, function and quality of life for the patient

SUMMARY:
Patients with total hip or knee replacement experiencing persistant problems are offered 3 weeks of intensive rehabilitation.

DETAILED DESCRIPTION:
Outcomes before, at the end of treatment and at 6 months follow up will be investigated. Data will be handled separately for the two groups of patients: 42 with a total hip replacement and 42 with a total knee replacement. Specific and generic outcomes will be collected.

ELIGIBILITY:
Inclusion Criteria:

- Patients with a total hip or knee replacement admitted for intensive rehabilitation

Exclusion Criteria:

* Patients unable to understand Danish
* Unable to participate in physical tests
* Unable to understand questionaires
* Unable to participate i 6 months follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have a total hip or knee replacement experiencing persistant problems, hence are admitted to a 3 week intensive rehabilitation period.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
HOOS/KOOS pain (0-100 score) | Change from baseline (0) to 3 weeks
  Hip or knee related pain
HOOS/KOOS ADL (0-100 score) | Change from baseline (0) to 3 weeks
  Hip or knee related activities of daily living
HOOS/KOOS quality of life (0-100 score) | Change from baseline (0) to 3 weeks
  Hip or knee related quality of life
HOOS/KOOS pain (0-100 score) | Change from 3 weeks to 7 months
  Hip or knee related pain
HOOS/KOOS ADL (0-100 score) | Change from 3 weeks to 7 months
  Hip or knee related activities of daily living
HOOS/KOOS quality of life (0-100 score) | Change from 3 weeks to 7 months
  Hip or knee related quality of life
Sit-to-stand test | Change from baseline (0) to 3 weeks
  Number of completed sit to stands in 30 seconds
Sit-to-stand test | Change from 3 weeks to 7 months
  Number of completed sit to stands in 30 seconds

SECONDARY OUTCOMES:
Patient acceptable symptom state (yes/no) | 3 weeks follow up
  Patients are asked with a single question if their current symptom state is acceptable
Patient acceptable symptom state (yes/no) | 7 months follow up
  Patients are asked with a single question if their current symptom state is acceptable
Pain catastrophising scale (0-52 score) | Baseline
  Current level of pain catastrophising with 0 being the best
Pain catastrophising scale (0-52 score) | 3 weeks
  Current level of pain catastrophising with 0 being the best
Pain catastrophising scale (0-52 score) | 7 months
  Current level of pain catastrophising with 0 being the best
Global rating of change (0-11 score) | Change from baseline to 3 weeks
  Likert scale where patients indicate their overall rating of change since the beginning of the intervention
Global rating of change (0-11 score) | Change from baseline to 7 months
  Likert scale where patients indicate their overall rating of change since the beginning of the intervention
The 5-level EQ-5D version (EQ-5D-5L) (0-5 scale) | Change from baseline (0) to 3 weeks
  EQ5D5L scores
The 5-level EQ-5D version (EQ-5D-5L) (0-5 scale) | Change from 3 weeks to 7 mothns
  EQ5D5L scores
EQ5D VAS (0-100 scale) | Change from baseline (0) to 3 weeks
  EQ5D Vas overall health
EQ5D VAS (0-100 scale) | Change from 3 weeks to 7 months
  EQ5D Vas overall health
HOOS/KOOS symptoms (0-100 score) | Change from baseline (0) to 3 weeks
  Hip or knee related symptoms
HOOS/KOOS symptoms (0-100 score) | Change from 3 weeks to 7 months
  Hip or knee symptoms
HOOS/KOOS sport/rec (0-100 score) | Change from baseline (0) to 3 weeks
  Hip or knee related sport/rec
HOOS/KOOS sport/rec (0-100 score) | Change from 3 weeks to 7 months
  Hip or knee related sport/rec
6 minute walk test | Change from baseline (0) to 3 weeks
  The distance a patient can walk in 6 minutes
6 minute walk test | Change from 3 weeks to 7 months
  The distance a patient can walk in 6 minutes
40 meter fast paced walk test | Change from baseline (0) to 3 weeks
  The time a patient uses walking 40 meters fast
40 meter fast paced walk test | Change from 3 weeks to 7 months
  The time a patient uses walking 40 meters fast
Stair test | Change from baseline (0) to 3 weeks
  The time a patient uses to ascend and decend a staircase
Stair test | Change from 3 weeks to 7 months
  The time a patient uses to ascend and decend a staircase

OTHER OUTCOMES:
Patient acceptable symptom state (yes/no) | Baseline
  Patients are asked with a single question if their current symptom state is acceptable
Employment status (yes/no/part time) | Baseline
Employment status (yes/no/part time) | 7 months

CONTACTS AND LOCATIONS:
Locations (1):
- Horsens Regional Hospital, Brædstrup, Denmark

IPD SHARING:
Plan to Share IPD: Undecided